CLINICAL TRIAL: NCT03332368
Title: Clinical Study on Prevention and Treatment of Recurrent and Metastasis of Triple Negative Breast Cancer(TNBC) With Traditional Chinese Medicine(TCM)
Brief Title: Clinical Study on Triple Negative Breast Cancer With Chinese Medicine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheng Liu (Other)
Responsible Party: Sponsor-Investigator, Sheng Liu, Principal Investigator, Clinical Professor, Longhua Hospital
Organization: Longhua Hospital (Other)
Other Study IDs: LonghuaH(TNBC); Special Research on TCM (Other: State Administration of Traditional Chinese Medicine)
Record Dates: First submitted 2017-10-24; First posted 2017-11-06 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Progression-Free-Survival; Recurrence; Overall Survival
Keywords: Triple-negative breast cancer; Traditional Chinese Medicine
MeSH Terms: conditions — Recurrence; Triple Negative Breast Neoplasms | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TCM exposure group: TCM exposure group were treated with traditional Chinese medicine while the other do not treated with that
  Interventions: Other: Traditional Chinese medicine

INTERVENTIONS:
Other: Traditional Chinese medicine — Chinese medicine has a long history of prevention and treatment of breast cancer, the effect is obvious. Chinese medicine its mechanism of action is from the whole, adjust the body yin and yang, blood, viscera function balance, emphasizing the combination of governance and external treatment of the combination of thinking, according to different clinical syndromes, using syndrome differentiation.

SUMMARY:
Breast cancer is one of the most serious threat to women's health of malignant tumors, also the most common causes of cancer death in women.Triple-negative breast cancer (TNBC) refers to the immunohistochemical detection of estrogen receptor (ER), progesterone receptor (PR), human epidermal growth factor receptor-2 (Her-2) are negative.Compared with other types of breast cancer, TNBC has a high degree of invasion,local recurrence and metastasis. Also,TNBC can not use endocrine therapy and lack of molecular targeting for Her-2 target therapy.Meanwhile other biological agents are too expensive,so the current clinical therapy only can use in China is chemotherapy,the average survival time is about 2 years.

Fortunately,due to the impact of traditional Chinese medicine(TCM) in China, the majority of breast cancer patients have received varying degrees of TCM treatment, and because of TNBC patients can not be more mature endocrine therapy and anti-molecular targeted therapy Benefits, Chinese medicine play an important role in TNBC patients.TCM regulate immune function, inhibit tumor growth, Anti-recurrence and metastasis, to extend the survival of patients with tumor, and relative to chemotherapy drugs and molecular targeted drugs,improve the quality of life.In addition ,comparing with the biological agents,Chinese medicine prices are relatively low,and can be worth using widely.

With the development of evidence-based medicine, and gradually recognize the importance of comprehensive treatment of breast cancer, Cancer Treatment Model has been proposed,.That is, to take Chinese medicine, surgery, radiotherapy and chemotherapy, endocrine therapy and biological immunization and other standardized, individualized comprehensive treatment. The introduction of evidence-based medicine into the field of research, will be beneficial to the objective evaluation of TCM syndrome differentiation in the treatment of refractory breast cancer in the characteristics and advantages in order to promote the use of.

This study based on TCM syndrome differentiation and treatment, and adopts multi-center, randomized, double-blind and controlled research methods to evaluate whether the intervention of traditional Chinese medicine can improve the TNBC patients with disease-free survival (DFS), overall survival(OS),and the best time to intervene in traditional Chinese medicine; also the establishment of the exact effect, obvious advantages and evidence, can be promoted in line with clinical practice of the program, the formation of refractory breast Cancer and Western medicine combined with clinical path, and relying on the national clinical research base of Chinese medicine information platform, the construction of clinical information management cloud platform, the formation of active medical service process, the establishment of refractory breast cancer combined with clinical prevention and treatment center, improve the life quality level of TNBC patients.

The study contains 5 locations,including Longhua Hospital, Shuguang Hospital,Yueyang Hospital,Zhejiang Traditional Chinese Medicine Hospital and Fudan University Cancer Hospital.Considering of the results of the study at MD Anderson Cancer Center in foreign countries showed that the 3-year survival rate of TNBC patients was significantly shorter than that of non-TNBC patients (74% vs.89%, P <0.01) To be at least 10% survival rate.At the same time, considering the case lost rate of 20%, calculated by PASS software, the number of samples for each group of 310 cases, a total of 620 cases of cohort study. According to whether to take traditional Chinese medicine,all the participants are divided into exposure group and non-exposure group, the number of observations per group is 310.

Before the research, all participants needs to fill in the informed consent form, investigators introduce the clinical research related matters to them and record the basic situation. The Chinese medicine exposure group take Chinese medicine(San Yin Decoction ) besides of original Western medicine , non-exposed group only received Western medicine treatment, a total of two years.All results are recorded in the CRF table,and use SPSS18.0, Stata10.0 and other statistical software for data to analysis.

ELIGIBILITY:
Participants' inclusion criteria are as follows:

1. The primary breast cancer after surgical treatment, the pathological diagnosis of breast epithelial tumors (breast cancer), ER, PR and Her-2 immunohistochemical results were negative;
2. no recurrence of metastasis;
3. card score ≥ 60 points;
4. Female patients aged 18-75 years (including 18,75 years);
5. there is no serious organic or functional disorders, no drugs and food allergy;
6. willing to receive treatment, observation and inspection.

Participants' exclusion criteria are as follow:

1. does not meet the inclusion criteria;
2. patients expected to survive <6 months;
3. combined with cardiovascular and cerebrovascular, liver, kidney, hematopoietic system of serious primary disease and mental illness;
4. breastfeeding, pregnancy or women preparing for pregnancy;
5. allergies and allergies to a variety of drugs;
6. are participating in other drug subjects.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Reference to the 《Chinese Medical Association prepared the "clinical treatment guidelines • tumor volume"》， all postoperative cases have been clearly diagnosed as triple negative breast cancer by pathological cells and immunohistochemistry.
Sampling Method: Non-Probability Sample
Enrollment: 620 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival, PFS | 2 years
  Progression-Free-Survival (PFS): Calculates the time from patient treatment to disease recurrence or death due to disease progression.Unit: month
Overall Survival，OS | 2 years
  Overall Survival (OS) refers to the time from the beginning of treatment to death due to any cause.Unit: month

SECONDARY OUTCOMES:
TCM Symptom Scale | 2 years
  CM Symptom: basing on the "Chinese Medicine New Drug Clinical Research Guidelines (Trial)" (China Medical Science and Technology Press, 2002) ,the investigators evaluate the TCM Symptom every 3 months,and using scoring method to evaluate efficacy.All results are recorded in the CRF table.
  Significant improvement: the integral value after treatment than the integral value before treatment decreased by ≥ 70% Partial improvement: the integral value after treatment than the integral value before treatment decreased by ≥ 30%; No improvement: before and after treatment without change or after treatment integral value than the integral value before treatment decreased by <30%
Karnofsky Performance Status（KPS） | 2 years
  The Karnofsky Performance Status (KPS) ranking runs from 100 to 0, where 100 is "perfect" health and 0 is death. Practitioners occasionally assign performance scores in between standard intervals of 10. The investigators evaluate the KPS score every 3 months,and using scoring method to evaluate efficacy.All results are recorded in the CRF table.
  Improved: KPS score increased> 10 points and maintained for more than 4 weeks; Stable: KPS score no significant change; Worsening: KPS score reduced by <10 points
ECOG score | 2 years
  he Eastern Cooperative Oncology Group (ECOG) score (published by Oken et al. in 1982), runs from 0 to 5, with 0 denoting perfect health and 5 death,The investigators evaluate the KPS score every 3 months,and using scoring method to evaluate efficacy.All results are recorded in the CRF table.
European Organization for Research and Treatment of Cancer (EORTC) Breast-Cancer-Specific Quality of Life Questionnaire (EORTC QLQ-BR23) | 2 years
  his questionnaire is focus on participants' physical condition and the quality of life .The investigators evaluate the score every 3 months,and using scoring method to evaluate efficacy.All results are recorded in the CRF table.

OTHER OUTCOMES:
Clinical indicators | 2 years
  his includes Tumor markers,immune function evaluation,chest CT/MRI and Abdominal B-ultrasound in order to monitor whether there is the tumor recurrence and metastasis.All the participants do Tumor markers check and immune function evaluation every 3 months,also chest CT/MRI and scan their bone every 6 months.
Adverse Event | 2 years
  By setting up safety indicators to assess drug safety and whether the participants have any adverse reactions. All the participants need to check Blood, urine, feces,also liver and kidney function,Abdominal B-ultrasound,Electrocardiogram every 3 months.If the investigators find any adverse events, they need to assess the event according to the WHO acute and subacute side effects of the performance and indexing criteria for assessment, divided into 0,1,2,3,4.All results are recorded in the CRF table.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Sheng, Master, Study Chair — Longhua Hospital; Qin Yuenong, Master, Study Director — Longhua Hospital
Locations (5):
- China (5):
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Longhua Hosptial, Shanghai, Shanghai Municipality
  - ShuGuang Hospital, Shanghai, Shanghai Municipality
  - Yueyang Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Traditional Chinese Medicine Hospital, Zhejiang, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen J, Qin Y, Sun C, Hao W, Zhang S, Wang Y, Chen J, Chen L, Ruan Y, Liu S. Clinical study on postoperative triple-negative breast cancer with Chinese medicine: Study protocol for an observational cohort trial. Medicine (Baltimore). 2018 Jun;97(25):e11061. doi: 10.1097/MD.0000000000011061. PMID 29923998